CLINICAL TRIAL: NCT01206907
Title: AN OPEN-LABEL, NON-RANDOMIZED, MULTICENTER EFFECTIVENESS, SAFETY AND TOLERABILITY STUDY OF OXYMORPHONE HCl IMMEDIATE-RELEASE ORAL LIQUID IN OPIOID-TOLERANT PEDIATRIC SUBJECTS WITH CHRONIC PAIN REQUIRING AN AROUND THE CLOCK OPIOID
Brief Title: Effectiveness, Safety, and Tolerability Study of Oxymorphone Immediate Release (IR) Oral Liquid in Opioid Tolerant Pediatric Subjects
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study is no longer required for the PREA for this product.
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director CR & D, Endo Pharmaceuticals, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3319-301
Record Dates: First submitted 2010-09-17; First posted 2010-09-22 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Pain
Keywords: sickle cell anemia; juvenile rheumatoid arthritis; burn victim; cancer; Chronic pain of malignant or non-malignant etiology
MeSH Terms: conditions — Chronic Pain; Anemia, Sickle Cell; Arthritis, Juvenile; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: oxymorphone IR — oxymorphone IR liquid

SUMMARY:
The purpose of this study is to evaluate the effectiveness, tolerability, and safety of oxymorphone immediate release (IR) oral liquid as an analgesic in pediatric subjects having severe to moderate chronic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 2 to ≤6 years of age, inclusive
2. Chronic cancer or non-cancer pain, currently requiring treatment of pain with a strong opioid for at least 5 days (3 of 5 days at a dose >1 mg/kg qd oral morphine equivalent)
3. Expected to continue to require a strong opioid for pain relief for at least 4 months
4. Able to swallow the oxymorphone HCl immediate-release oral liquid
5. Have been informed of the nature of the study and informed consent and assent by minor (if IRB required) has been obtained from the legally responsible parent/legal guardian in accordance with IRB requirements

Exclusion Criteria:

1. Known allergy to, or a significant reaction to, oxymorphone or another opioid
2. Life expectancy <4 months
3. Any clinical condition in the investigator's opinion that would preclude participation
4. Plan to undergo a surgical procedure within 1 month of study entry or anytime during study
5. Currently prescribed a long-acting opioid (eg., Kadian® morphine sulfate extended release) as part of their analgesic regimen
6. Received any investigational medication within 30 days prior to the first dose of study medication, or are scheduled to receive an investigational drug other than oxymorphone during the course of the study
7. An ileostomy
8. Received a monoamine oxidase inhibitor (MAOI) within 14 days prior to the start of study medication
9. Investigator anticipates that the subject would be unable to comply with the protocol
10. Parent/legal guardian is unable to complete the subject's daily study medication diary
11. Parent/legal guardian is unable to effectively communicate the subject's status to the investigator

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity from baseline to last assessment using the Face, Legs, Activity, Cry, Consolability (FLACC) pain scale. | weekly for 1 month during titration
Change in pain intensity from baseline to last assessment using the Face, Legs, Activity, Cry, Consolability (FLACC) pain scale. | bi-weekly for three months in the maintenance phase

SECONDARY OUTCOMES:
Safety Assessment of Adverse Events, vital signs including oxygen saturation, Blood Pressure, and Heart Rate. | weekly for 1 month during titration
Safety Assessment of Adverse Events, vital signs including oxygen saturation, Blood Pressure, and Heart Rate. | bi-weekly for 3 months in the maintenance phase